CLINICAL TRIAL: NCT05587790
Title: EMPOWER Weight Loss Program for Obesity in Rural and Underserved Areas Pilot Study
Brief Title: EMPOWER Rural Extension Weight Management Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22642
Record Dates: First submitted 2022-07-18; First posted 2022-10-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: Obesity; Overweight; Weight Loss; Rural; Nonmetropolitan; Protein; Fiber
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: Before and after study design with one interventional group and no control or placebo group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Weight Management Intervention (Experimental): During a 12-month period, participants will attend a total of 17 diet improvement sessions, each of which will last approximately 45-minutes. Twelve sessions will be held in the first 5 months and will be focused on safe and efficient weight loss. The participants will learn to create a personalized weight loss diet from their kitchen based on their diet practice and food preference. The next 10 sessions will be held in the last 7 months and will be focused on weight maintenance and healthy eating. The participants will build skills to select foods and create meals that prevent them from overeating. Flexibility in session completion will be allowed to accommodate busy schedules, vacation, and potential internet access challenges.
  Interventions: Behavioral: Weight Management Intervention

INTERVENTIONS:
Behavioral: Weight Management Intervention — Participants attend virtual dietary education sessions and over time create a diet plan that satisfies their individual needs. Participants aim to lose 1-2 pounds weekly until a BMI of 25 is reached. Participants are evaluated through daily self-weighing, dietary records, and anthropometric measures of waist and hip circumference, and body composition.

SUMMARY:
This research is to expand a virtual weight loss and weight maintenance program to rural counties of Illinois. The program uses dietary and lifestyle modifications for adults with obesity. The EMPOWER weight loss program has proven to be effective in 3 previous trials. In this research, we target a rural participant population. Individuals in rural locations are more likely to be affected by obesity and have unique barriers to weight loss related to geographic isolation including access to health care, preventative care, grocery stores, social networks, internet, and cell service.

DETAILED DESCRIPTION:
EMPOWER is a remote weight management program that uses an online textbook platform, E-Text, and mobile web application, MealPlot. This pilot study will test for feasibility of the EMPOWER program in a rural population prior to launching a full-scale study. Acceptability measurements will be collected at 3 months to evaluate for needed changes; Participants of the pilot study will be permitted to continue on with the full program.

EMPOWER is a 1-year intervention. Data is collected via 24-hour record and daily weighing using a Wi-Fi-enabled scale. 24-hour records and daily weights are collected within the program's proprietary MealPlot website. EMPOWER consists of 17 online sessions (45 minutes/each) and 12 individual advising sessions with a nutrition coach.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* BMI in overweight to above range;
* not currently pregnant or lactating;
* willing to access Wi-Fi via home or free public Wi-Fi location at least once a week for 45 minutes
* access to a working email
* willing to weigh daily and provide data either via Bluetooth, Wi-Fi, or manual input
* willing to lose 20 lb. or more and maintain a healthy weight for one year thereafter;
* Continue daily-weighing for 12-months after the year-long intervention (Daily weigh for a total of 2 years);
* fluent in reading and writing English.
* live within one of the counties of the covered Extension Education offices: Eastern (Clark, Crawford, Edgar), Northern (Jo Daviess, Stephenson, Winnebago), Western (Macoupin, Christian, Jersey, Montgomery)

Exclusion Criteria:

* age <18 or >75 years;
* severe chronic diseases;
* underweight to normal BMI;
* currently pregnant;
* currently lactating;
* failed to commit to daily weighing;
* failed to submit 3, 24 hour records;
* underwent bariatric surgery or planning on having bariatric surgery within the next year including: Roux-en-Y Gastric Bypass, Sleeve Gastrectomy, Duodenal Jejunal Bypass with Sleeve Gastrectomy, Duodenal Switch, Laparoscopic Adjustable Gastric Banding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Enrollment | 3 Months
  Achieving target enrollment 16
Retention | 3 Months
  Successful retention dropout <20% (13/16)
Completion of eText | 12 Months
  Completion of eText (75% completion)
Completion of study measures | 12 Months
  Completion of 80% of study measures (24-hour records, in-person anthropometric testing)
Acceptability | 3 Months
  4/5 on average for all program components and overall program using Likert scales (ranging 1-5) of acceptability (comprehensive program, MealPlot, eText, nutrition coaching) collected via survey.

SECONDARY OUTCOMES:
Weight loss | 1 Year
  Change in weight
Dietary habits - protein density | 1 Year
  protein density change from baseline to 12 months.
Dietary Habits - fiber density | 1 Year
  Fiber density change from baseline to 12 months.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UIUC Extension, Freeport, Illinois
  - UIUC Extension, Hillsboro, Illinois
  - UIUC Extension, Marshall, Illinois

IPD SHARING:
Plan to Share IPD: No
All researchers must pass Core Human Subjects training through CITI. Confidentiality of data collected will be maintained by assigning each participant a three-digit identification (ID) code which will be used to enter all data in an electronic database. ID codes will be used on all documents and materials as the only form of identification; no names will be used. All files and participant documentation will be stored in locked filing cabinets. Electronic documents, forms and data will be stored in a Health Data folder on Box. Only the primary investigator, co-investigator, and research team will have access to stored data.
  Any data collected via email will be completed using ID codes and deleted and emptied from trash following data collection. The primary investigator will immediately destroy documents that are obtained from individuals who do not qualify for the study, as determined during the pre-screening and screening steps. These documents will be shredded.